CLINICAL TRIAL: NCT00324571
Title: A Randomized, Open Label, Parallel Design Study of Renagel® Phosphate Binder Versus Calcium-Based Phosphate Binders in Hemodialysis Patients
Brief Title: Dialysis Clinical Outcomes Revisited (DCOR) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTC-68-401
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer

INTERVENTIONS:
Drug: Sevelamer hydrochloride
Drug: Calcium-based phosphate binder

SUMMARY:
This is a randomized, open-label, parallel-design study to be conducted at 75 centers within the United States. The study will be described to hemodialysis patients. Informed consent will be obtained and the inclusion/exclusion criteria reviewed. Eligible patients will be randomized to receive either Renagel or a calcium-based binder.

Starting from the randomization date, mortality data including survival, death date and cause of death (vital status information) and morbidity data including hospitalization date will be recorded for all patients. These data will be collected until the end of the study (December 31, 2004, ± 2 weeks). Patients completing or terminating from the study will return to the phosphate binder prescribed by their usual healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* patients must be 18 years of age or older,
* on dialysis for more than 3 months,
* require phosphate binder therapy,
* have Medicare as their primary insurance.

Exclusion Criteria:

* dysphagia,
* swallowing disorders,
* severe gastrointestinal motility disorders,
* bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2001-03; Study Completion 2006-02

PRIMARY OUTCOMES:
Efficacy will be evaluated based on a comparison of the association of Renagel use versus calcium-based phosphate binder use on all-cause mortality, cause-specific mortality (cardiovascular, infection, other), and all-cause hospitalization.
Safety will be assessed based on an evaluation of related serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (73):
- United States (72):
  - Gambro Healthcare-Gadsden, Gadsden, Alabama
  - nTouch Research, Huntsville, Alabama
  - Kidney Health Institute, LLC, Tucson, Arizona
  - Gambro Healthcare, El Cerrito, California
  - Palomar Medical Group, Escondido, California
  - Gambro Healthcare-Los Angeles, Los Angeles, California
  - Balboa Nephrology Medical Group, San Diego, California
  - Nephrology Educational Services and Research, Tarzana, California
  - Lowry Dialysis Center, Denver, Colorado
  - Nephrology Associates, P.C., Bridgeport, Connecticut
  - Gambro Healthcare-Hartford, Hartford, Connecticut
  - Nephrology Associates, New Britain, Connecticut
  - InterAmerican Dialysis, Coral Gables, Florida
  - DaVita Crystal River Dialysis, Crystal River, Florida
  - Gambro Healthcare-Miami, Miami, Florida
  - Miami Kidney Group, Miami, Florida
  - Pensacola Nephrology, P.A., Pensacola, Florida
  - Gambro Healthcare-Plantation, Plantation, Florida
  - America Dialysis, St. Petersburg, Florida
  - Genesis Clinical Research Corp, Tampa, Florida
  - Gambro Healthcare-Americus, Americus, Georgia
  - nTouch Research, Atlanta, Georgia
  - Gambro Healthcare-Douglas, Douglas, Georgia
  - Gambro Healthcare-Douglasville, Douglasville, Georgia
  - Dublin Nephrology, Dublin, Georgia
  - Georgia Kidney Associates, Inc., Marietta, Georgia
  - Gambro Healthcare-Rome, Rome, Georgia
  - Gambro Healthcare-Savannah, Savannah, Georgia
  - MacNeal Renal Lifeline Services, Berwyn, Illinois
  - Southwest Nephrology, Evergreen Park, Illinois
  - Horizon Healthcare Associates, Olympia Fields, Illinois
  - Renal Care Associates, S.C., Peoria, Illinois
  - Gambro Healthcare-Springfield Central, Springfield, Illinois
  - Lincolnland Dialysis, Springfield, Illinois
  - Nephrology Specialists, PC., Valparaiso, Indiana
  - Wichita Dialysis Center East, Wichita, Kansas
  - Wichita Nephrology, Wichita, Kansas
  - Northwest Louisiana Nephrology, LLC., Shreveport, Louisiana
  - BMA of Washington, Bethesda, Maryland
  - Gambro Healthcare-Frederick, Frederick, Maryland
  - Associates in Nephrology, P.C., Brockton, Massachusetts
  - Western New England Renal and Transplant Associates, Inc., Springfield, Massachusetts
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Nephrology Associates, P.C., Columbus, Mississippi
  - University of Missouri-Kansas City, Kansas City, Missouri
  - DaVita Crystal City Dialysis, St Louis, Missouri
  - Nephrology and Endocrine Associates, Las Vegas, Nevada
  - Bronx Westchester Medical Group, The Bronx, New York
  - Mountain Kidney Associates, P.A., Asheville, North Carolina
  - nTouch Research, Raleigh, North Carolina
  - Wake Nephrology/Wake Dialysis Clinic, Raleigh, North Carolina
  - Gambro Healthcare-Wilson, Wilson, North Carolina
  - Kidney and Hypertension Center, Cincinnati, Ohio
  - Ohio State University College of Pharmacy, Columbus, Ohio
  - FMC of Bethlehem, Allentown, Pennsylvania
  - Fresenius Medical Care, Greensburg, Pennsylvania
  - Hypertension and Kidney Specialists, Lancaster, Pennsylvania
  - DaVita Lewistown Dialysis Center, Lewistown, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - P.C. & Associates, Philadelphia, Pennsylvania
  - Nesbitt College of Pharmacy and Nursing Department of Pharmacy Practice, Wilkes-Barre, Pennsylvania
  - Gambro Healthcare-Aiken, Aiken, South Carolina
  - Midsouth Nephrology Consultants, Memphis, Tennessee
  - Dallas Nephrology Associates, Dallas, Texas
  - Nephrology, Dialysis and Transplant Association, Houston, Texas
  - West Houston Dialysis, Houston, Texas
  - San Antonio Kidney Disease Center, San Antonio, Texas
  - Gambro Healthcare - Charlottesville, Charlottesville, Virginia
  - Clinical Research and Consulting Center, LLC, Fairfax, Virginia
  - Clinical Research of Tidewater, Norfolk, Virginia
  - Virginia Commonwealth University, Division of Nephrology, Richmond, Virginia
  - Vancouver Clinic Inc., P.S., Vancouver, Washington
- Clinical Las Americas, San Juan, Puerto Rico

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086